CLINICAL TRIAL: NCT07038265
Title: Patient-centered Cardiac rehaBilitation pRogramE in Post Acute Coronary Syndrome:Identification of Key Barriers and Evaluation of Personalized Intervention (BREAK-trial)
Brief Title: Patient-centered Personalized Cardiac Rehabilitation in Post Acute Coronary Syndrome (BREAK-trial)
Acronym: BREAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut d'Investigació Biomèdica de Bellvitge (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Fundació La Marató de TV3 (Other)
Responsible Party: Principal Investigator, Cristina Enjuanes Grau, Coordinator of Community Heart Failure Unit, Cardiology Department. MD, PhD, Institut d'Investigació Biomèdica de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: IDIBELL- 202309 10; 202309 10 (Other Grant/Funding Number: Fundació La Marató 2022)
Record Dates: First submitted 2025-04-04; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Acute Coronary Syndromes (ACS); Cardiac Rehabilitation; Frailty; Women; Women's Health
Keywords: frailty; sarcopenia; cardiac rehabilitation; gender perspective; acute coronary syndrome; coronary artery disease; patient-centered care
MeSH Terms: conditions — Acute Coronary Syndrome; Frailty; Sarcopenia; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Patients will be recruited during 14 months, and will be followed for a fixed period of 6 months. The study protocol will be approved by the institutional review boards of the center (Bellvitge Biomedical Research Institute, IDIBELL).
  The trial will be designed and implemented by the BREAK Steering Committee. Oversight of the study will be conducted by the Chair and the two Co-Chairs in liason with the BREAK Executive Committee. Safety will be reported by local investigators in accordance with the current legislation that regulates pharmacovigilance in Spain.
  End-point evaluation of the primary outcome will be performed by an independent end-point committee blinded to the group allocation of patients.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Usual cardiac rehabilitation program
  Interventions: Other: Usual Care
- Personalized intervention program (Experimental): BREAK intervention group with more alternatives of aerobic and strength exercises and also offering remote options for fragile patients
  Interventions: Behavioral: Personalised treatment

INTERVENTIONS:
Behavioral: Personalised treatment — Patients going through a personalized intervention program
  Arms: Personalized intervention program
Other: Usual Care — Usual cardiac rehabilitation program
  Arms: Standard of care

SUMMARY:
The primary objective of this study is to compare an integrated, multidisciplinar patient-centered CRP (Cardiac Rehabilitation Program) (intervention group) especially focused on covering the needs for the female and fragile population to the usual care conventional CRP (control group)

DETAILED DESCRIPTION:
The Break-CR study is designed as an unicentric, open, randomized controlled trial, blind end-point evaluation and adjudication, to compare the feasibility, efficacy, and safety of a patient-centered CR-program versus usual care in patients after an acute coronary syndrome (ACS). The project aims to identify these barriers and design a CR-intervention to overcome said barriers and evaluate its usefulness in clinical practice.

The first part of this study consists of a qualitative study to specifically determine barriers, difficulties and facilitators that condition the participation of women in the CRPs, the second part of the study is undertaken to address the underrepresentation of women in CRPs and provide a solution to the recognized need to redesign CR programs to respond to the unique physiological and psychosocial needs of women. The aim is to design a groundbreaking intervention model that will respond to this need because it will incorporate all the factors on which a CR programme should be based, from a woman's perspective, from the beginning to the end, while also adressing the needs of the fragile portion ACS survivors.

It is hypothesized that the Break-CR program would be able to demonstrate greater improvements in incorporation and adherence of women and fragile patients to CR-programs, enhanced functional benefits, as well as improve patient-satisfaction and quality of life. Finally, the fundamental purpose is to enhance poor health outcomes of women and fragile patients with coronary diseases and to provide a solution that will contribute to bridge the health gap that exists in the field of cardiovascular diseases in health systems.

ELIGIBILITY:
Inclusion Criteria:

1. Patient aged ≥ 18 years
2. Patients discharged within the last 30 days after an admission for ACS or in the discharge planning process for an admission for ACS.
3. The patient is able to fully communicate with the research team and comply with all study procedures.
4. The patient voluntarily signs and dates the informed consent form approved by the ethics committee

Exclusion Criteria:

1. Age <18 years
2. Participation in another clinical trial
3. Moderate or severe cognitive impairment in the absence of a competent caregiver
4. Absence of social support
5. Institutionalized patient
6. Life expectancy <1 year
7. Candidates for end-of-life care
8. Severe psychiatric illness
9. Planned cardiac surgery including transplant or circulatory support implant
10. Death before hospital discharge in patients included in the hospital discharge planning phase
11. Carrier of heart transplant.
12. Patient unable or refusing to give written informed consent to participate
13. Patients who, in the opinion of the investigator, are unsuitable candidates for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Estimated)
Dates: Start 2025-05-26 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Improvement in functional capacity | First visit and 3 months after hospital discharge (after completing rehabilitation program)
  The primary endpoint of the study will be a composite functional capacity score, designed to capture the overall improvement in cardiorespiratory fitness following the rehabilitation intervention.
  This composite score will integrate the standardized change (from baseline to the end of the intervention) in the following four variables:
  1. Peak oxygen uptake (VO₂ peak, in ml/kg/min), measured via cardiopulmonary exercise testing (CPET).
  2. Six-minute walk distance (6MWD, in meters), assessed using the six-minute walk test.
  3. Maximal metabolic equivalents (METs), achieved during CPET.
  4. Exercise test duration (in minutes), defined as the total time sustained during the treadmill or cycle ergometer test under a standardized, symptom-limited protocol.
  Each of these variables will be converted to z-scores based on the distribution of change scores in the study population. The composite score will be calculated as the mean of the four standardized values

SECONDARY OUTCOMES:
Physical Activity. IPAQ | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital discharge
  Adherence to physical activity will be evaluated with the International Physical Activity Questionnaire (IPAQ). The IPAQ classifies individuals into three categories of physical activity level based on intensity, frequency, and total energy expenditure (measured in MET·minutes/week):
  Category 1: Low Physical Activity:
  The person does not meet the criteria for moderate or high physical activity.
  Considered sedentary or insufficiently active.
  Category 2: Moderate Physical Activity. A person meets any of the following:
  * 3 days/week of vigorous activity ≥20 minutes/day, or
  * 5 days/week of moderate activity and/or walking ≥30 minutes/day, or
  * 5 days/week of any combination of walking, moderate, or vigorous activity totaling ≥600 MET·minutes/week.
  Category 3: High Physical Activity. A person meets either:
  * 3 days/week of vigorous activity accumulating ≥1,500 MET·minutes/week, or
  * 7 days/week of any combination of walking, moderate or vigorous activity totaling ≥3,000 MET·minutes/week
Physical Activity. Podometer | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital dischargeFirst visit and 6 months after hospital discharge
  According to pedometer readings which will be given to patients (steps/day), physical activity is categorized as follows:
  Sedentary or inactive < 5,000 steps/day Low active 5,000-9,999 steps/day Active 10,000-12,499 steps/day Very active ≥ 12,500 steps/day
Psychological status | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital dischargeFirst Visit and 6 months after hospital discharge
  Psychological status will be evaluated for screening of anxiety and depression (PHQ-9 and GAD-7 scales).
  The PHQ-9 is a 9-item questionnaire used to screen for depression. Each item is scored from 0 (not at all) to 3 (nearly every day), with a total score range of 0-27. Cut-off points:
  5-9: mild depression 10-14: moderate depression 15-19: moderately severe depression 20-27: severe depression
  The GAD-7 is a 7-item scale assessing generalized anxiety. Each item is scored 0-3 (same as PHQ-9), total score range: 0-21. Cut-off points:
  5-9: mild anxiety 10-14: moderate anxiety 15-21: severe anxiety
  A score ≥10 on either scale suggests clinically relevant symptoms, warranting further evaluation.
Dietary Changes | In-hospital evaluation and 6 months after hospital discharge
  ChatGPT Plus To assess dietary changes, we will use two validated tools: the DEBQ (Dutch Eating Behavior Questionnaire) and the PREDIMED Mediterranean Diet questionnaire.
  The DEBQ evaluates emotional, external, and restrained eating behaviors using 33 items rated on a 5-point scale (from "never" to "very often"). It helps identify if a patient eats more in response to emotions, sensory cues, or dieting efforts. Higher scores in each subscale indicate a stronger influence of that behavior on eating patterns.
  The PREDIMED questionnaire has 14 questions and measures adherence to the Mediterranean diet. Each healthy habit (e.g., using olive oil, eating fruits/vegetables, low processed food intake) scores 1 point.
  Scores ≥9 = good adherence, <9 = low adherence.
  These tools allow monitoring of diet quality and behavior-related eating changes
Body composition | First visit and 3 months after hospital discharge (after completing rehabilitation program)
  Nutritional status will be evaluated with the use of bioimpedanciometry (BIA), monitoring changes in body composition such as % of muscle and fat mass.
Sarcopenia | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital discharge
  Sarcopenia will be assessed in patients using handgrip dynamometry, expressed in kilograms (kg). Handgrip strength (HGS) is a validated proxy for overall muscle strength and is widely used in clinical settings for sarcopenia screening. According to the international norms published by Tomkinson et al. (2025), cut-off values will be based on sex- and age-specific percentiles.
  Patients with HGS values below the 20th percentile for their age and sex will be considered at risk of sarcopenia. This threshold aligns with evidence suggesting that the lowest quintile is predictive of poorer health outcomes and increased mortality. These percentiles provide a robust, standardized reference to guide early intervention.
Frailty | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital discharge
  Frailty will be assessed using the Short Physical Performance Battery (SPPB), a validated tool that evaluates lower extremity function through three components:
  Balance (side-by-side, semi-tandem, tandem stand)
  Gait speed (usual pace over 4 meters)
  Chair stands (time to rise from a chair five times)
  Each component is scored from 0 to 4, giving a total score range of 0 to 12 (higher scores = better function).
  Cut-off points for frailty classification:
  0-6 points: frail
  7-9 points: pre-frail
  10-12 points: robust
  This tool helps identify patients at risk of mobility disability and adverse outcomes and is recommended for use in both research and clinical practice.
Patient reported quality of life | First visit and 3 months after hospital discharge (after completing rehabilitation program)
  Changes in quality of life will be assessed using two validated instruments: the EuroQol-5D (EQ-5D) and the HeartQoL (HRQoL) questionnaire.
  (EQ-5D)
  This tool evaluates health across 5 dimensions:
  Mobility Self-care Usual activities Pain/discomfort Anxiety/depression
  Each dimension has 3 levels: no problems, some problems, and extreme problems. It also includes a visual analogue scale (VAS) from 0 (worst imaginable health) to 100 (best imaginable health), allowing patients to rate their overall health state. Higher scores indicate better perceived health.
  HRQoL
  The HRQoL is a disease-specific questionnaire for patients with ischemic heart disease. It has 14 items divided into two dimensions:
  Physical (10 items) Emotional (4 items)
  Each item is scored from 0 (worst HRQoL) to 3 (best HRQoL). Scores are averaged for each subscale and the global score; higher scores reflect better quality of life. Changes over time can reflect improvements or deterioration in health perception
Sleep quality | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital discharge
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index (PSQI), a standardized questionnaire that evaluates sleep patterns over the past month.
  The PSQI consists of 19 self-rated items grouped into 7 components:
  Subjective sleep quality Sleep latency Sleep duration Habitual sleep efficiency Sleep disturbances Use of sleeping medication Daytime dysfunction
  Each component is scored from 0 to 3, producing a global score ranging from 0 to 21.
  Scores ≤5: good sleep quality Scores >5: poor sleep quality
  Higher scores reflect worse sleep quality. The PSQI is widely used in both research and clinical practice to monitor sleep-related changes and identify individuals with potential sleep disorders.
Sexual dysfunction | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital discharge
  Sexual dysfunction will be assessed using validated, sex-specific questionnaires:
  For men: IIEF (International Index of Erectile Function)
  The IIEF evaluates male sexual function over the past 4 weeks using 15 items distributed across 5 domains:
  Erectile function (items 1-5, 15) Orgasmic function (items 9-10) Sexual desire (items 11-12) Intercourse satisfaction (items 6-8) Overall satisfaction (items 13-14)
  Each item is scored from 0 or 1 to 5, with higher scores indicating better sexual function.
  Erectile dysfunction is usually classified as:
  1-10: severe 11-16: moderate 17-25: mild to moderate 26-30: normal
  For women: FSM (Female Sexual Function Questionnaire)
  This tool consists of 19 items grouped into 6 domains:
  Desire (items 1-2) Arousal (items 3-6) Lubrication (items 7-10) Orgasm (items 11-13) Satisfaction (items 14-16) Pain (items 17-19)
  Some items are reverse-scored (8, 10, 12, 17-19). Higher total and subscale scores indicate better sexual function.
Readmission and mortality rates | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital discharge
  Readmission Rate (All-Cause and Cardiovascular)
  Patient outcomes will include evaluation of hospital readmissions, classified as:
  All-cause readmissions: any reason for hospital admission after discharge. Cardiovascular readmissions: admissions due to heart-related conditions (e.g., heart failure, myocardial infarction, arrhythmia).
  We will register both the rate (percentage of patients readmitted) and the total number of readmissions. A lower readmission rate reflects better clinical stability and care continuity.
  Mortality (All-Cause and Cardiovascular)
  Mortality will be monitored and classified into:
  All-cause mortality: death from any origin. Cardiovascular mortality: death due to cardiac or vascular causes (e.g., sudden cardiac death, stroke, heart failure).
  These indicators will evaluate patient prognosis and treatment effectiveness over the follow-up period.
Adherence to program | First visit; 3 months after discharge (after completing rehabilitation program)
  Patient adherence and retention will be evaluated as follows:
  1.1 Adherence analysis: the total percentage of exercise sessions attended in both groups (conventional vs domiciliary program). And also adherence to the different types of sessions (respiratory, relaxation, aerobic and strength) 1.2. Retention rate: the number of participants who finish the training divided by the number of randomized patients.
Patient experience | First visit; 3 months (after completing rehabilitation program) and 6 months after hospital discharge
  Patient's experience with both the cardiac rehabilitation program and the use of technology will be assessed using a LIKERT scale (1 Not at all to 5 A lot) asking the following questions:
  * How do you think a cardiac rehabilitation program can impact your health?
  * How do you think the use of information technology can impact your health?
  The results will be analyzed before starting the program and at the end to determine if patient's impression has changed.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Enjuanes, MD, PhD, Principal Investigator — Institut d'Investigació Biomèdica de Bellvitge
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No